CLINICAL TRIAL: NCT00537407
Title: An Open-label, Randomized, 5-arm, Parallel-group Study of the Effects on Viral Kinetics, Safety and Pharmacokinetics of Different Dosing Regimens of Debio 025 in Combination With Peginterferon Alpha-2a and Ribavirin in Chronic HCV Genotype 1 Patients Who Are Non Responders to Standard Peginterferon Alpha and Ribavirin Treatment
Brief Title: A Study of Debio 025 in Combination With PegIFN Alpha-2a and Ribavirin in Chronic HCV Patients Non-responders to Standard Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 025-HCV-207; DEB025A2207 (Other: Sponsor Code)
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis; Hepatitis C | interventions — alisporivir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment Arm A (Experimental): Debio 025 (alisporivir) 400 mg orally once daily + peg-IFNα2a 180 μg subcutaneously (sc) once weekly + ribavirin 1000 or 1200 mg/day orally for 29 days followed by peg-IFNα2a 180 μg sc once weekly + ribavirin 1000 or 1200 mg/day orally administered for 44 or 68 weeks depending upon response
  Interventions: Drug: Debio 025; Drug: Peg-IFNα2a; Drug: Ribavirin
- Treatment Arm B (Experimental): Debio 025 (alisporivir) 400 mg orally once daily for 29 days followed by peg-IFNα2a 180 μg sc once weekly + ribavirin 1000 or 1200 mg/day orally administered for 44 or 68 weeks depending upon response
  Interventions: Drug: Debio 025; Drug: Peg-IFNα2a; Drug: Ribavirin
- Treatment Arm C (Experimental): Debio 025 (alisporivir) 400 mg orally once daily + peg-IFNα2a 180 μg sc once weekly for 29 days followed by peg-IFNα2a 180 μg sc once weekly + ribavirin 1000 or 1200 mg/day orally administered for 44 or 68 weeks depending upon response
  Interventions: Drug: Debio 025; Drug: Peg-IFNα2a; Drug: Ribavirin
- Treatment Arm D (Experimental): Debio 025 (alisporivir) 800 mg orally once daily + peg-IFNα2a 180 μg sc once weekly + ribavirin 1000 or 1200 mg/day orally for 29 days followed by peg-IFNα2a 180 μg sc once weekly + ribavirin 1000 or 1200 mg/day orally administered for 44 or 68 weeks depending upon response
  Interventions: Drug: Debio 025; Drug: Peg-IFNα2a; Drug: Ribavirin
- Treatment Arm E (Experimental): Debio 025 (alisporivir) orally at a loading dose of 400 mg twice daily for 7 days followed by 400 mg/day for 22 days + peg-IFNα2a 180 μg sc once weekly + ribavirin 1000 or 1200 mg/day orally for 29 days followed by peg-IFNα2a 180 μg sc once weekly + ribavirin 1000 or 1200 mg/day orally administered for 44 or 68 weeks depending upon response
  Interventions: Drug: Debio 025; Drug: Peg-IFNα2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Debio 025 — Debio 025 supplied as a 100 mg/mL oral solution
  Other Names: Alisporivir
Drug: Peg-IFNα2a — Peg-IFNa2a supplied in 180 μg/0.5 mL prefilled syringes
  Other Names: PEGASYS
Drug: Ribavirin — Ribavirin supplied as 200 mg tablets
  Other Names: Copegus

SUMMARY:
Debio 025 (alisporivir) is an oral cyclophilin inhibitor with a new mechanism of action demonstrating potent anti-hepatitis C virus (HCV) activity in pre-clinical models and patients.

The current standard of care (SOC) in HCV patients consists of a combination of peg-IFN alpha and ribavirin. Treatment duration and ribavirin dose depend on the genotype treated. Only 40-50% of patients with genotype 1 achieve a sustained viral response (SVR). This study assesses whether Debio 025 administered in combination with peg-IFN alpha 2a and ribavirin can improve the outcome of treatment in this group of patients.

DETAILED DESCRIPTION:
This is a multicentre, open-label, randomized, 5 arm parallel-group, multiple dose study in 50 chronic hepatitis C virus (HCV) genotype 1 non-responders to standard treatment with peg-IFN alpha (2a or 2b) and ribavirin. The entire study lasts a maximum of 96 weeks and consists of a 48- or 72-week treatment period (according to response). A follow-up visit to assess the sustained viral response (SVR) takes place 24 weeks after treatment cessation, i.e., at study Week 72 or 96, or earlier for discontinued study participants.

There were 2 parts in the treatment period. Part 1 lasted from Day 1 to Day 29 (Weeks 1 to 4); Part 2 lasted from Week 5 to Week 48 or 72.

During Part 1 of treatment (Weeks 1 to 4), participants are randomized to 1 of 5 treatment arms and receive 4 weeks of Debio 025 (alisporivir) monotherapy, Debio 025 combined with standard dose peg-IFNα2a, or 1 of 3 triple therapies combining different doses of Debio 025 with peg-IFNα2a and ribavirin at standard doses.

During Part 2 of treatment (Weeks 5 to 48 or 72), participants receive standard doses of peg-IFNα2a/ribavirin dual therapy for 44 or 68 weeks, depending on their response to treatment. At Week 12, participants who do not achieve ≥ 2 log10 decrease in HCV RNA are withdrawn and considered treatment failures. Participants who have undetectable HCV RNA levels and/or ≥ 2 log10 decrease in HCV RNA continue treatment until Week 24. At Week 24, participants who still have detectable HCV RNA levels are withdrawn and considered treatment failures. Participants with undetectable HCV RNA levels at Weeks 12 and 24 continue treatment until Week 48. At Week 24, "slow responders" (defined as participants with a detectable, but > 2 log10 decrease in HCV RNA levels at Week 12 and undetectable levels at Week 24) are eligible to continue treatment until Week 72.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 60 years of age.
* Hepatitis B negative and human immunodeficiency virus (HIV) negative.
* Diagnosed with hepatitis C genotype I and not responsive to treatments such as peginterferon alpha-2a or 2b and ribavirin for at least 12 weeks.
* Adequate liver function (Child-Pugh-Turcotte score A) and other laboratory parameters within acceptable range.
* Females may participate only if they cannot become pregnant, i.e., are surgically sterile, post-menopausal, or using 2 reliable contraceptive methods.
* Male patients must be surgically sterile or utilizing a barrier contraceptive method.
* For female patients of child bearing potential, negative pregnancy test within 1 week of first investigational product administration.

Exclusion Criteria:

* Treatment with any investigational drug within 6 months prior to the start of the study.
* Ongoing or recent use of antiviral medication within 1 month before the start of the study.
* A known bad reaction or intolerance to Debio 025, peginterferon alpha-2a, and/or ribavirin.
* Presence or history of any severe related disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raf Crabbé, MD, Study Director — Debiopharm International S.A.
Locations (7):
- United States (7):
  - Scripps Clinic Liver Disease Research Center, La Jolla, California
  - University of Florida, Gainesville, Florida
  - University of Miami Center for Liver Diseases, Miami, Florida
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Methodist Transplant Physicians, Dallas, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Virginia Mason Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Part 1 Weeks 1-4
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D | Treatment Arm E
Started | 10 | 9 | 11 | 10 | 10
Completed | 10 | 9 | 11 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2 Weeks 5-48 or 72
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D | Treatment Arm E
Started | 10 | 9 | 11 | 10 | 10
Completed | 2 | 1 | 2 | 4 | 3
Not Completed | 8 | 8 | 9 | 6 | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants with at least a Baseline and 1 on- or post-treatment hepatitis C virus RNA assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D | Treatment Arm E | Total
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 10 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 11 | 10 | 10 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (6.62) | 52.6 (5.94) | 49.9 (10.71) | 48.5 (9.87) | 52.8 (6.51) | 51.0 (8.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 5 | 3 | 21
  Male | 7 | 4 | 6 | 5 | 7 | 29
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 11 | 10 | 10 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in log10 Hepatitis C Virus RNA at Day 29 in the Debio 025 Triple Therapy Treatment Arms (A, D, and E)
Description: Hepatitis C virus RNA was quantified in plasma samples using real time polymerase chain reaction.
Time Frame: Baseline to Day 29
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Log10(IU/mL)
Arm/Group | Treatment Arm A | Treatment Arm D | Treatment Arm E
Number analyzed (Participants) | 10 | 10 | 10
Log10(IU/mL) | -0.881 (1.0099) | -2.321 (1.4644) | -2.020 (1.4031)

2. Secondary Outcome: Change From Baseline in log10 Hepatitis C Virus RNA at Day 29 in the Debio 025 Monotherapy and Dual Therapy Treatment Arms (B and C)
Description: Hepatitis C virus RNA was quantified in plasma samples using real time polymerase chain reaction.
Time Frame: Baseline to Day 29
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Log10(IU/mL)
Arm/Group | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 9 | 11
Log10(IU/mL) | 0.285 (0.3273) | -0.608 (0.7558)

3. Secondary Outcome: log10 Hepatitis C Virus RNA at Day 29
Description: Hepatitis C virus RNA was quantified in plasma samples using real time polymerase chain reaction.
Time Frame: Day 29
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Log10(IU/mL)
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D | Treatment Arm E
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 10
Log10(IU/mL) | 5.567 (1.0165) | 6.662 (0.3295) | 5.827 (0.7270) | 4.000 (1.4325) | 4.245 (1.6337)

4. Secondary Outcome: Percentage of Participants With a Rapid Viral Response at Day 29
Description: A participant had a rapid viral response if their viral RNA was undetectable (< 10 IU/mL).
Time Frame: Day 29
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D | Treatment Arm E
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 10
percentage of participants | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 28.5] | 10 [0.3 to 44.5] | 10 [0.3 to 44.5]

5. Secondary Outcome: Percentage of Participants With an Early Viral Response at Week 12
Description: A participant had an early viral response if their viral RNA had decreased ≥ 2 log10 at Week 12 compared to Baseline.
Time Frame: Baseline to Week 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D | Treatment Arm E
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 10
percentage of participants | 30.0 | 11.1 | 27.3 | 70.0 | 30.0

6. Secondary Outcome: Percentage of Participants With an End-of-treatment Response at the End of Treatment (Week 48 or 72)
Description: A participant had an end-of-treatment response if their viral RNA was undetectable (< 10 IU/mL).
Time Frame: End of treatment (Week 48 or 72)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D | Treatment Arm E
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 10
percentage of participants | 20.0 | 11.1 | 18.2 | 10.0 | 30.0

7. Secondary Outcome: Percentage of Participants With a Sustained Viral Response 24 Weeks After the End of Treatment (Week 72 or 96)
Description: A participant had a sustained viral response if their viral RNA was undetectable (< 10 IU/mL).
Time Frame: 24 weeks after the end of treatment (Week 72 or 96)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D | Treatment Arm E
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 10
percentage of participants | 0.0 | 0.0 | 9.1 | 0.0 | 10.0

ADVERSE EVENTS:
Time Frame: Within 72 weeks
Description: Safety population: All participants who received any dose of Debio 025 and had at least 1 post-baseline assessment.
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D | Treatment Arm E
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 1/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9 | 11/11 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A (N=10) | Treatment Arm B (N=9) | Treatment Arm C (N=11) | Treatment Arm D (N=10) | Treatment Arm E (N=10)
Acute Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A (N=10) | Treatment Arm B (N=9) | Treatment Arm C (N=11) | Treatment Arm D (N=10) | Treatment Arm E (N=10)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 4 (4) | 1 (1) | 4 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aphthous Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Faecal Volume Increased (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces Pale (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hunger (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (3) | 3 (3) | 3 (5)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensitivity of Teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Early Satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 2 (2) | 4 (4) | 5 (5) | 8 (10)
Influenza Like Illness (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection Site Haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Irritability (General disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Local swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 3 (5)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail bed infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bacteria urine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Blood Triglycerides Increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase Increased (Investigations) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mean cell volume increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteocalcin Increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine Output Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Resorption Bone Increased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 2 (2) | 2 (2) | 6 (8) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychomotor Hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Depressed Mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 4 (4) | 5 (5) | 0 (0)
Memory impairment (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Glycosurea (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation Irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspneoa (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (3)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 2 (2)
Rash Macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin Odour Abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Venous insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other